CLINICAL TRIAL: NCT00441740
Title: Vinorelbine and Gemcitabine Versus Docetaxel and Gemcitabine as First Line Treatment in Patients With Advanced or Metastatic Non Small Cell Lung Cancer (NSCLC). A Prospective , Multicenter, Randomized, Phase III Trial
Brief Title: Randomized Trial With Vinorelbine and Gemcitabine Versus Docetaxel and Gemcitabine in Patients With Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hellenic Oncology Research Group (Other)
Collaborators: University Hospital of Crete (Other)
Responsible Party: V.Georgoulias, Hellenic Oncology Research Group
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT/04.04
Record Dates: First submitted 2007-02-28; First posted 2007-03-01 (Estimated); Last update posted 2008-10-31 (Estimated); Status verified 2008-10

CONDITIONS: Non Small Cell Lung Cancer
Keywords: NSCLC; 1st line treatment; Gemcitabine; Vinorelbine; Docetaxel
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Vinorelbine; Gemcitabine; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): VG
  Interventions: Drug: Vinorelbine; Drug: Gemcitabine
- 2 (Experimental): DG
  Interventions: Drug: Docetaxel; Drug: Gemcitabine

INTERVENTIONS:
Drug: Vinorelbine — Vinorelbine (oral) 70 mg/m2, on days 1 and 15 every 4 weeks for 6 cycles
  Other Names: Navelbine
  Arms: 1
Drug: Gemcitabine — Gemcitabine 900 mg/m2 on days 1 and 15 every 4 weeks for 6 cycles
  Other Names: Gemzar
  Arms: 1
Drug: Docetaxel — Docetaxel 75 mg/m2 intravenous on day 8 every 3 weeks for 6 cycles
  Other Names: Taxotere
  Arms: 2
Drug: Gemcitabine — Gemcitabine 1000 mg/m2 intravenous, on days 1 and 8 every 3 weeks for 6 cycles
  Other Names: Gemzar
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate whether the gemcitabine/vinorelbine combination versus the gemcitabine/docetaxel combination as first line treatment, offers a survival advantage in patients with locally advanced/metastatic NSCLC.

DETAILED DESCRIPTION:
Cisplatin-based chemotherapy represented the backbone of treatment of advanced NSCLC. However, several trials comparing platinum versus non-platinum based chemotherapy regimens failed to demonstrate a statistically significant difference in terms of time to tumor progression or survival. Newer agents such as gemcitabine, docetaxel and vinorelbine have shown significant activity in the treatment of NSCLC. Gemcitabine/vinorelbine combination as first line treatment has demonstrated a response rate (RR) of 18-43% and a median overall survival (OS) of 9.8-13 months. Similarly, the gemcitabine/docetaxel combination has shown a RR 32-35% and a median OS of 9-12 months. Given their proven efficacy, the combination of these two doublets, would be interesting.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed, unresectable locally advanced (stage IIIB with pleural effusion) and/or metastatic (stage IV) NSCLC
* No previous therapy for advanced/metastatic NSCLC is allowed
* Age > 18 years
* Bidimensionally measurable disease
* Performance status (WHO) 0-2
* Adequate liver (serum bilirubin < 1.5 times the upper normal limit (UNL); AST and ALT < 2.5 times the UNL in the absence of demonstrable liver metastases, or < 5 times the UNL in the presence of liver metastases); adequate renal function (serum creatinine < 1.5 times the UNL); and bone marrow (neutrophils ≥ 1.5x 109 /L, and platelets ≥ 100x 109 /L) function
* Previous radiotherapy, either in the adjuvant setting or for the treatment of metastatic disease is allowed provided that the measurable lesions are outside the radiation fields
* Life expectancy of more than 3 months
* Patient able to take oral medication
* At least 4 weeks since prior radiotherapy
* Written informed consent

Exclusion Criteria:

* Active infection
* History of significant cardiac disease (unstable angina, congestive heart failure, myocardial infarction within the previous 6 months, ventricular arrhythmias)
* Malnutrition (loss of ≥ 20% of the original body weight)
* Performance status: 3-4
* Sensor or motor neuropathy > grade I
* Second primary malignancy, except for non-melanoma skin cancer
* Psychiatric illness or social situation that would preclude study compliance
* Pregnant or lactating women
* Known, symptomatic central nervous system metastases

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 419 (Actual)
Dates: Start 2004-04; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Overall survival | 1 year

SECONDARY OUTCOMES:
Response rate | Objective responses confirmed by CT or MRI (on 3rd and 6th cycle)
Time to tumor progression | 1 year
Toxicity | Toxicity assessment on each chemotherapy cycle
Quality of life | Assessment every two cycles

CONTACTS AND LOCATIONS:
Overall Officials: Vassilis Georgoulias, MD, Principal Investigator — University Hospital of Crete, Dep of Medical Oncology
Locations (9):
- Greece (9):
  - University General Hospital of Alexandroupolis, Dep of Medical Oncology, Alexandroupoli
  - " General Hospital, 1st, 3rd, 8th Dep of Pulmonary Diseases, Athens
  - "Laikon" General Hospital, Medical Oncology Unit, Propedeutic Dep of Internal Medicine, Athens
  - "Metaxa's" Anticancer Hospital of Piraeus,1st Dep of Medical Oncology, Athens
  - 401 Military Hospital, Medical Oncology Unit, Athens
  - Air Forces Military Hospital, Dep of Medical Oncology, Athens
  - IASO" General Hospital of Athens, 1st Dep of Medical Oncology, Athens
  - Sismanogleio General Hospital, 1st, 2nd Dep of Pulmonary Diseases, Athens
  - "Theagenion" Anticancer Hospital of Thessaloniki, Thessaloniki